CLINICAL TRIAL: NCT02911532
Title: Tissue Engineering Conjunctiva Transplantation and Conjunctival Sac Formation for the Treatment of Pterygium and Atretoblepharia
Brief Title: Tissue Engineering Conjunctiva for the Treatment of Pterygium and Atretoblepharia
Acronym: TECTPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160816
Record Dates: First submitted 2016-08-26; First posted 2016-09-22 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Pterygium
Keywords: pterygium; tissue engineering; atretoblepharia
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optical Coherence tomography (Experimental)
  Interventions: Procedure: Tissue engineering conjunctiva transplantation

INTERVENTIONS:
Procedure: Tissue engineering conjunctiva transplantation — During the operation,transplant the tissue engineering conjunctiva to the conjunctiva loss position

SUMMARY:
The purpose of this study is to determine whether tissue engineering conjunctiva is effective in the treatment of pterygium and atretoblepharia.

DETAILED DESCRIPTION:
The most important area for research on the pterygium are the recurrence occurred after operation. Now the best way to prevent the recurrence is autologous conjunctival stem cell transplantation, but this way of operation can cause lack of conjunctiva and conjunctival scar, even may effect the later glaucoma surgery. For the atretoblepharia patients, amniotic membrane transplantation and autologous oral mucosa transplantation can not make effect to alleviate it. In this pilot project, investigators would like to study the effect of tissue engineering conjunctiva transplantation in the treatment of pterygium and tissue engineering conjunctiva transplantation combined with conjunctiva sac formation for the treatment of atretoblepharia. This will allow us to determine if useful data can be obtained, and if so, lead to further studies in various conjunctiva loss caused by trauma, infections, and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Primary and recurrent pterygium patients,atretoblepharia patients
2. Voluntarily signed informed consent
3. No surgery and anesthesia contraindications.

Exclusion Criteria:

1. The patients combined systemic diseases
2. Reject study and follow visit
3. Patients don't accept the tissue engineering conjunctiva
4. Cannot tolerate surgery or anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
The epithelial defect size of the transplanted tissue engineering conjunctiva | the 7 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Weiyun Shi, sponsor, Study Chair — director of shandong eye hospital
Locations (1):
- Shandong Eye Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Varssano D, Shalev H, Lazar M, Fischer N. Pterygium excision with conjunctival autograft: true survival rate statistics. Cornea. 2013 Sep;32(9):1243-50. doi: 10.1097/ICO.0b013e31828ce09c. PMID 23594771
- [Background] Mahar PS, Manzar N. The study of etiological and demographic characteristics of pterygium recurrence: a consecutive case series study from Pakistan. Int Ophthalmol. 2014 Feb;34(1):69-74. doi: 10.1007/s10792-013-9797-4. Epub 2013 Jun 18. PMID 23775605
- [Background] Farid M, Pirnazar JR. Pterygium recurrence after excision with conjunctival autograft: a comparison of fibrin tissue adhesive to absorbable sutures. Cornea. 2009 Jan;28(1):43-5. doi: 10.1097/ICO.0b013e318183a362. PMID 19092404
- [Background] Kaufman SC, Jacobs DS, Lee WB, Deng SX, Rosenblatt MI, Shtein RM. Options and adjuvants in surgery for pterygium: a report by the American Academy of Ophthalmology. Ophthalmology. 2013 Jan;120(1):201-8. doi: 10.1016/j.ophtha.2012.06.066. Epub 2012 Oct 11. PMID 23062647
- [Background] Tan DT, Chee SP, Dear KB, Lim AS. Effect of pterygium morphology on pterygium recurrence in a controlled trial comparing conjunctival autografting with bare sclera excision. Arch Ophthalmol. 1997 Oct;115(10):1235-40. doi: 10.1001/archopht.1997.01100160405001. PMID 9338666
- [Background] Sandra S, Zeljka J, Zeljka VA, Kristian S, Ivana A. The influence of pterygium morphology on fibrin glue conjunctival autografting pterygium surgery. Int Ophthalmol. 2014 Feb;34(1):75-9. doi: 10.1007/s10792-013-9799-2. Epub 2013 Jun 4. PMID 23733279
- [Background] Hirst LW, Sebban A, Chant D. Pterygium recurrence time. Ophthalmology. 1994 Apr;101(4):755-8. doi: 10.1016/s0161-6420(94)31270-x. PMID 8152771
- [Background] Ozer A, Yildirim N, Erol N, Yurdakul S. Long-term results of bare sclera, limbal-conjunctival autograft and amniotic membrane graft techniques in primary pterygium excisions. Ophthalmologica. 2009;223(4):269-73. doi: 10.1159/000210444. Epub 2009 Apr 2. PMID 19339811
- [Background] Zheng K, Cai J, Jhanji V, Chen H. Comparison of pterygium recurrence rates after limbal conjunctival autograft transplantation and other techniques: meta-analysis. Cornea. 2012 Dec;31(12):1422-7. doi: 10.1097/ICO.0b013e31823cbecb. PMID 22643650
- [Background] Hirst LW. The treatment of pterygium. Surv Ophthalmol. 2003 Mar-Apr;48(2):145-80. doi: 10.1016/s0039-6257(02)00463-0. PMID 12686302
- [Background] Li M, Zhu M, Yu Y, Gong L, Zhao N, Robitaille MJ. Comparison of conjunctival autograft transplantation and amniotic membrane transplantation for pterygium: a meta-analysis. Graefes Arch Clin Exp Ophthalmol. 2012 Mar;250(3):375-81. doi: 10.1007/s00417-011-1820-8. Epub 2011 Sep 21. PMID 21935607
- [Background] Hirst LW. Recurrence and complications after 1,000 surgeries using pterygium extended removal followed by extended conjunctival transplant. Ophthalmology. 2012 Nov;119(11):2205-10. doi: 10.1016/j.ophtha.2012.06.021. Epub 2012 Aug 11. PMID 22892149
- [Background] Gris O, Guell JL, del Campo Z. Limbal-conjunctival autograft transplantation for the treatment of recurrent pterygium. Ophthalmology. 2000 Feb;107(2):270-3. doi: 10.1016/s0161-6420(99)00041-x. PMID 10690823